CLINICAL TRIAL: NCT05209217
Title: Open Study of the Neurobiological Effects of Intranasal Ketamine in Children and Adults With Bipolar Disorder - Fear of Harm Phenotype
Brief Title: Open Study of the Neurobiological Effects of Intranasal Ketamine in Children and Adults With Bipolar Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mclean Hospital (Other)
Collaborators: Juvenile Bipolar Research Foundation (Other)
Responsible Party: Principal Investigator, Martin H Teicher, Director of the Developmental Biopsychiatry Research Program, Mclean Hospital
Other Study IDs: 2017P001822
Record Dates: First submitted 2018-10-26; First posted 2022-01-26 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant Group: Participants will all have history of good to excellent clinical response to intranasal ketamine for at least two months and on a treatment schedule varying from use every other day to every fifth day. Participants will be tested one or two days beyond their customary administration date and again 2-3 hours after their administration of ketamine.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Intranasal administration of their customary prescribed dose

SUMMARY:
Aim 1: Test the hypothesis that participants with Bipolar Disorder - Fear of Harm Phenotype have an enhanced amygdala fMRI response to fearful threatening stimuli, increased resting beta and gamma EEG spectral activity in temporal leads and blunted posterior insula response to cold when partially withdrawn from ketamine with normalization of these responses following intranasal administration of ketamine.

Aim 2. Test the hypothesis that ketamine alters response to fearful-threatening visual stimuli and cold sensation by altering functional connectivity of the amygdala and insula with the hypothalamus, thalamus, hippocampus and ventromedial prefrontal cortex, and identify specific alterations that correlate with degree of pre-post ketamine change.

Aim 3. Test the hypothesis that low-dose medicinal ketamine, unlike high-dose recreation ketamine, is not associated with an increase in number of focal areas of abnormality on morphometric scans based on duration of use.

DETAILED DESCRIPTION:
Clinically, the Fear of Harm phenotype is characterized by early age of onset, severe mood swings, treatment resistance, separation anxiety, fearful-aggressive obsessions, parasomnias (e.g. night-terrors) and thermal dysregulation (Papolos et al. 2009). These youth typically received little benefit from standard treatments (i.e., antipsychotic medication and mood stabilizers) often wind up home-schooled due to excessive fears of the school environment and frequently require multiple periods of inpatient care (Papolos et al. 2009; Papolos et al. 2013). Key features seen in FOH that distinguish these youths from other youths with BD include fear sensitization and thermal dysregulation. Children with FOH often experience thermal discomfort (e.g., feeling hot, excessive sweating) in neutral ambient temperature conditions, as well as no discomfort during exposure to the cold, and alternate noticeably between being excessively hot in the evening and cold in the morning (Murphy, Frei, and Papolos 2014). Ketamine, an NMDA receptor antagonist was selected as a potential treatment for FOH because of its effectiveness in the reduction of fear sensitization and capacity to dose-dependently lower body temperature in animal studies, and has been found to be clinically efficacious in the treatment of FOH (Papolos et al. 2018; Papolos et al. 2013). There are two main reasons for proposing to conduct a neuroimaging study. First, intranasal ketamine can produce an almost immediate improvement in clinical state. This makes it possible to scan a subject whose dose of ketamine has largely worn off in order to assess blood flow and functional connectivity and then to rescan the individual within hours of receiving intranasal ketamine in order to correlate degree of clinical improvement with alterations in blood flow and connectivity. This will provide information on both the neurobiological basis of ketamine response and information on the possible biological underpinnings of FOH. Second, there is some concern, based on a report of examining brain scans in chronic ketamine abusers, that ketamine in daily doses 10X higher than clinically prescribed every 3-4 days can produce some evidence for structural brain damage4. Hence, it would be valuable to scan individuals undergoing long term treatment with intranasal ketamine to rule out or monitor for pathological changes in brain structure.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age 14 - 40 years
* Clinical diagnosis of Bipolar Disorder -Fear of Harm Phenotype
* Meets Papolos criteria for FOH based on independent interviews.
* Taking intranasal ketamine for at least 2 months.
* Must be on an every three or every four-day dosing regimen
* Dosage will not exceed 300 mg per dosing interval.
* Willing to delay ketamine dose by 2 days past their prescribed dosing interval
* Prior experience having tolerated this degree of delay.
* Willing to participate in daily assessments during period of ketamine withdrawal prior to traveling to Belmont ,MA.
* Willing to provide urine sample to screen for drugs of abuse (all participants and pregnancy in females.)

Exclusion Criteria:

* Any psychiatric hospitalization within the past 6 months
* Lifetime history of suicide attempts
* Co-occurring substance use disorders
* Any change in concomitant medications within the last 2 months

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Total sample size will be 20 subjects, with approximately equal number of males and females.
  Subjects recruited for the study will be between 14-40-years-of-age who meet DSM-5 criteria for Bipolar Disorder, Papolos criteria for FOH Phenotype, have been taking intranasal ketamine for at least two months
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
BOLD fMRI response in amygdala | Prior to and 2-3 hours following ketamine administration
  Change in BOLD measured by functional Magnetic Resonance Imaging (fMRI) to images of threatening versus neutral facial expressions.
BOLD fMRI response in posterior insula | Prior to and 2-3 hours following ketamine administration
  Correlation between BOLD measured by functional Magnetic Resonance Imaging (fMRI) and degree of cold stimulation of non-dominant hand.

SECONDARY OUTCOMES:
Functional connectivity between amygdala and insula | Prior to and 2-3 hours following ketamine administration
  Seed-to-seed and seed-to-voxel functional connectivity analysis of rs-fMRI data.
EEG spectral activity measures | Prior to and 2-3 hours following ketamine administration
  Absolute and relative power in low beta (15-26), high beta (28-40), low gamma (42-53) and high gamma (55-67) frequency bands using 32-channel Electrical Geodesics, Inc. EEG.
Profile of Mood State (POMS) scale. | Prior to and 2-3 hours following ketamine administration
  Ratings of tension and total mood score on the POMS.

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Teicher, MD, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share with other researchers

REFERENCES:
- [Background] Alsop DC, Detre JA, Golay X, Gunther M, Hendrikse J, Hernandez-Garcia L, Lu H, MacIntosh BJ, Parkes LM, Smits M, van Osch MJ, Wang DJ, Wong EC, Zaharchuk G. Recommended implementation of arterial spin-labeled perfusion MRI for clinical applications: A consensus of the ISMRM perfusion study group and the European consortium for ASL in dementia. Magn Reson Med. 2015 Jan;73(1):102-16. doi: 10.1002/mrm.25197. Epub 2014 Apr 8. PMID 24715426
- [Background] Anderson IM, Juhasz G, Thomas E, Downey D, McKie S, Deakin JF, Elliott R. The effect of acute citalopram on face emotion processing in remitted depression: a pharmacoMRI study. Eur Neuropsychopharmacol. 2011 Jan;21(1):140-8. doi: 10.1016/j.euroneuro.2010.06.008. PMID 20599362
- [Background] Castellanos FX, Margulies DS, Kelly C, Uddin LQ, Ghaffari M, Kirsch A, Shaw D, Shehzad Z, Di Martino A, Biswal B, Sonuga-Barke EJ, Rotrosen J, Adler LA, Milham MP. Cingulate-precuneus interactions: a new locus of dysfunction in adult attention-deficit/hyperactivity disorder. Biol Psychiatry. 2008 Feb 1;63(3):332-7. doi: 10.1016/j.biopsych.2007.06.025. Epub 2007 Sep 21. PMID 17888409
- [Background] Craig AD, Bushnell MC. The thermal grill illusion: unmasking the burn of cold pain. Science. 1994 Jul 8;265(5169):252-5. doi: 10.1126/science.8023144.
- [Background] Craig AD, Chen K, Bandy D, Reiman EM. Thermosensory activation of insular cortex. Nat Neurosci. 2000 Feb;3(2):184-90. doi: 10.1038/72131. PMID 10649575
- [Background] Craig AD, Reiman EM, Evans A, Bushnell MC. Functional imaging of an illusion of pain. Nature. 1996 Nov 21;384(6606):258-60. doi: 10.1038/384258a0. PMID 8918874
- [Background] Ding X, Ding J, Hua B, Xiong X, Xiao L, Peng F, Chen L, Pan X, Wang Q. Abnormal cortical functional activity in patients with ischemic white matter lesions: A resting-state functional magnetic resonance imaging study. Neurosci Lett. 2017 Mar 22;644:10-17. doi: 10.1016/j.neulet.2017.02.015. Epub 2017 Feb 9. PMID 28189742
- [Background] Fahim I, Ismail M, Osman OH. Role of 5-hydroxytryptamine in ketamine-induced hypothermia in the rat. Br J Pharmacol. 1973 Aug;48(4):570-6. doi: 10.1111/j.1476-5381.1973.tb08243.x. PMID 4274691
- [Background] Frankenstein UN, Richter W, McIntyre MC, Remy F. Distraction modulates anterior cingulate gyrus activations during the cold pressor test. Neuroimage. 2001 Oct;14(4):827-36. doi: 10.1006/nimg.2001.0883. PMID 11554801
- [Background] Heuchert, J. P., & McNair, D. M. (2012). Profile of Mood States, 2nd Edition (POMS-2). North Tonawanda, NY: Multi-Health Systems.
- [Background] Jenkinson M, Bannister P, Brady M, Smith S. Improved optimization for the robust and accurate linear registration and motion correction of brain images. Neuroimage. 2002 Oct;17(2):825-41. doi: 10.1016/s1053-8119(02)91132-8. PMID 12377157
- [Background] Kaufman, J., Birmaher, B., Axelson, D., Perepletchikova, F., Brent, D., & Ryan, N. (2016). Schedule for Affective Disorders and Schizophrenia for School Aged Children (6-18 Years). Kiddie-SADS - Lifetime Version (K-SADS-PL DSM-5 November 2016)
- [Background] La Cesa S, Tinelli E, Toschi N, Di Stefano G, Collorone S, Aceti A, Francia A, Cruccu G, Truini A, Caramia F. fMRI pain activation in the periaqueductal gray in healthy volunteers during the cold pressor test. Magn Reson Imaging. 2014 Apr;32(3):236-40. doi: 10.1016/j.mri.2013.12.003. Epub 2013 Dec 19. PMID 24468081
- [Background] Lapotka M, Ruz M, Salamanca Ballesteros A, Ocon Hernandez O. Cold pressor gel test: A safe alternative to the cold pressor test in fMRI. Magn Reson Med. 2017 Oct;78(4):1464-1468. doi: 10.1002/mrm.26529. Epub 2016 Oct 25. PMID 27779778
- [Background] Margulies DS, Kelly AM, Uddin LQ, Biswal BB, Castellanos FX, Milham MP. Mapping the functional connectivity of anterior cingulate cortex. Neuroimage. 2007 Aug 15;37(2):579-88. doi: 10.1016/j.neuroimage.2007.05.019. Epub 2007 May 24. PMID 17604651
- [Background] Murphy PJ, Frei MG, Papolos D. Alterations in skin temperature and sleep in the fear of harm phenotype of pediatric bipolar disorder. J Clin Med. 2014;3(3):959-71. doi: 10.3390/jcm3030959. PMID 25530872
- [Background] National Institute of Mental Health, N. (1985). CGI (Clinical Global Impression) Scale-NIMH. Psychopharmacol Bull, 12, 839-844.
- [Background] Papolos D, Frei M, Rossignol D, Mattis S, Hernandez-Garcia LC, Teicher MH. Clinical experience using intranasal ketamine in the longitudinal treatment of juvenile bipolar disorder with fear of harm phenotype. J Affect Disord. 2018 Jan 1;225:545-551. doi: 10.1016/j.jad.2017.08.081. Epub 2017 Aug 30. PMID 28866299
- [Background] Papolos D, Hennen J, Cockerham M. Obsessive fears about harm to self or others and overt aggressive behaviors in youth diagnosed with juvenile-onset bipolar disorder. J Affect Disord. 2005 Dec;89(1-3):99-105. doi: 10.1016/j.jad.2005.08.005. Epub 2005 Sep 27. PMID 16194571
- [Background] Papolos D, Hennen J, Cockerham MS, Lachman H. A strategy for identifying phenotypic subtypes: concordance of symptom dimensions between sibling pairs who met screening criteria for a genetic linkage study of childhood-onset bipolar disorder using the Child Bipolar Questionnaire. J Affect Disord. 2007 Apr;99(1-3):27-36. doi: 10.1016/j.jad.2006.08.014. Epub 2006 Oct 16. PMID 17049378
- [Background] Papolos D, Mattis S, Golshan S, Molay F. Fear of harm, a possible phenotype of pediatric bipolar disorder: a dimensional approach to diagnosis for genotyping psychiatric syndromes. J Affect Disord. 2009 Nov;118(1-3):28-38. doi: 10.1016/j.jad.2009.06.016. Epub 2009 Jul 23. PMID 19631388
- [Background] Papolos DF, Teicher MH, Faedda GL, Murphy P, Mattis S. Clinical experience using intranasal ketamine in the treatment of pediatric bipolar disorder/fear of harm phenotype. J Affect Disord. 2013 May;147(1-3):431-6. doi: 10.1016/j.jad.2012.08.040. Epub 2012 Nov 30. PMID 23200737
- [Background] Smith SM. Fast robust automated brain extraction. Hum Brain Mapp. 2002 Nov;17(3):143-55. doi: 10.1002/hbm.10062. PMID 12391568
- [Background] Steen RG, Hamer RM, Lieberman JA. Measuring brain volume by MR imaging: impact of measurement precision and natural variation on sample size requirements. AJNR Am J Neuroradiol. 2007 Jun-Jul;28(6):1119-25. doi: 10.3174/ajnr.A0537. PMID 17569971
- [Background] Wang C, Zheng D, Xu J, Lam W, Yew DT. Brain damages in ketamine addicts as revealed by magnetic resonance imaging. Front Neuroanat. 2013 Jul 17;7:23. doi: 10.3389/fnana.2013.00023. eCollection 2013. PMID 23882190
- [Background] Wang DJ, Alger JR, Qiao JX, Gunther M, Pope WB, Saver JL, Salamon N, Liebeskind DS; UCLA Stroke Investigators. Multi-delay multi-parametric arterial spin-labeled perfusion MRI in acute ischemic stroke - Comparison with dynamic susceptibility contrast enhanced perfusion imaging. Neuroimage Clin. 2013 Jul 6;3:1-7. doi: 10.1016/j.nicl.2013.06.017. eCollection 2013. PMID 24159561
- [Background] Whitfield-Gabrieli S, Nieto-Castanon A. Conn: a functional connectivity toolbox for correlated and anticorrelated brain networks. Brain Connect. 2012;2(3):125-41. doi: 10.1089/brain.2012.0073. Epub 2012 Jul 19. PMID 22642651
- [Background] Williams LM, Liddell BJ, Kemp AH, Bryant RA, Meares RA, Peduto AS, Gordon E. Amygdala-prefrontal dissociation of subliminal and supraliminal fear. Hum Brain Mapp. 2006 Aug;27(8):652-61. doi: 10.1002/hbm.20208. PMID 16281289
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Zhang LM, Zhou WW, Ji YJ, Li Y, Zhao N, Chen HX, Xue R, Mei XG, Zhang YZ, Wang HL, Li YF. Anxiolytic effects of ketamine in animal models of posttraumatic stress disorder. Psychopharmacology (Berl). 2015 Feb;232(4):663-72. doi: 10.1007/s00213-014-3697-9. Epub 2014 Sep 18. PMID 25231918